CLINICAL TRIAL: NCT02750319
Title: A Randomized, Double-Blind, Controlled Trial of Combined Amiodarone and N-Acetylcysteine Versus Amiodarone Plus Placebo for the Prevention of Atrial Fibrillation in High Risk Patients Undergoing Thoracic Surgery
Brief Title: Amiodarone and N-Acetylcysteine or Amiodarone Alone for Preventing Atrial Fibrillation After Thoracic Surgery
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Washington University School of Medicine (Other); The Cleveland Clinic (Other); Vanderbilt University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-307
Record Dates: First submitted 2016-04-21; First posted 2016-04-25 (Estimated); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Thoracic Surgery; Atrial Fibrillation in High Risk Patients
Keywords: Amiodarone; N-Acetylcysteine; 16-307
MeSH Terms: interventions — Amiodarone; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amiodarone + Placebo (Placebo Comparator): Amiodarone loading: 150 mg IV in PACU over one hour, then 1.0 gm/24h x 2 + NAC loading matching placebo; 50 mg/kg IV in PACU over one hour, then 50 mg/kg/24h x 2 NAC matched placebo continuously for 48 hours.
  Interventions: Drug: Amiodarone; Drug: Placebo
- Amiodarone + N-Acetylcysteine (Experimental): Amiodarone loading: 150 mg IV in PACU over one hour, then 1.0 gm/24h x 2 + NAC loading: 50 mg/kg IV in PACU over one hour, then 50 mg/kg/24h x 2 and then continuously for 48 hours.
  Interventions: Drug: Amiodarone; Drug: N-Acetylcysteine

INTERVENTIONS:
Drug: Amiodarone
Drug: N-Acetylcysteine
  Arms: Amiodarone + N-Acetylcysteine
Drug: Placebo
  Arms: Amiodarone + Placebo

SUMMARY:
This trial will be comparing the combination of amiodarone and NAC (n=122) to amiodarone alone and NAC matched placebo (n=122) to determine the rates with which sustained (lasting >30 seconds) or clinically significant POAF is reduced in high risk patients within 7 days after major thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old scheduled for elective thoracic surgery (segmentectomy, lobectomy or bi-lobectomy, pneumonectomy or esophagectomy) and meeting one of the four following risk criteria:

  * 1. Female & BNP ≥ 25pg/ml (no age limit)
  * 2. Male gender <75 & BNP ≥ 25pg/ml
  * 3. Male- age ≥75 (No BNP limit)
  * 4. History of prior AF
* Patients in sinus rhythm.
* Patients with stable respiratory status (no respiratory distress).
* Patients capable of providing written, informed consent.

Exclusion Criteria:

* Patients scheduled for extrapleural pneumonectomy.
* Hemodynamically unstable patients (not in cardiogenic shock or having an acute MI).
* Patients with 2nd or 3rd degree atrioventricular (AV) block.
* Patients with hypersensitivity to amiodarone or NAC.
* Patients already taking class Ic or III antiarrhythmic drugs.
* Hepatic insufficiency (≤2 times the upper normal limit of transaminase levels).
* Renal insufficiency (creatinine ≥2.0 mg/dl).
* Known pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
rate of sustained (lasting >30 seconds) or clinically significant post-operative atrial fibrillation (POAF) | within 7 days since operation
  Atrial arrhythmias will be considered and defined as atrial fibrillation/flutter (AF) lasting great than 30 seconds and/or sustained supraventricular tachycardia (SVT) that are detected by continuous telemetry or that are clinically significant, requiring intervention and documented by 12-lead ECG by the clinical staff.

CONTACTS AND LOCATIONS:
Overall Officials: David Amar, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - University of Washington School of Medicine in St. Louis, St Louis, Missouri
  - Memorial Sloan Kettering Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent only), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre (Consent only), Rockville Centre, New York
  - Memorial Sloan Kettering Nassau (Consent only), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/